CLINICAL TRIAL: NCT00764699
Title: Effect of Increlex® on Children With Crohn Disease
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: PI left institution
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: Tercica (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB08-00213
Record Dates: First submitted 2008-10-01; First posted 2008-10-02 (Estimated); Results first posted 2018-03-02 (Actual); Last update posted 2018-03-02 (Actual); Status verified 2018-02

CONDITIONS: Crohn Disease
Keywords: poor growth; inflammatory bowel disease
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases | interventions — mecasermin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- rhIGF (Experimental): Treatment with rhIGF (Increlex)
  Interventions: Drug: rhIGF (Increlex)

INTERVENTIONS:
Drug: rhIGF (Increlex) — rhIGF will be administered as a subcutaneous injection per the following schema: First 2 weeks: 40 mcg/kg BID; Weeks 3 and 4: 80 mcg/kg BID; Subsequent weeks: 120 mcg/kg BID.
  Other Names: Increlex

SUMMARY:
Patients with Crohn disease often have poor weight gain and short stature, yet the etiology of the poor growth is not well defined. Studies in chronically ill patients who do not have Crohn disease have suggested that inflammation causes IGF-1 deficiency due to inadequate IGF-1 generation. Previous studies of GH use in Crohn patients have demonstrated improvement in linear growth, weight and bone mineralization. However, GH can cause glucose intolerance in chronically ill children, particularly those who require treatment with corticosteroids. Recently the FDA has approved recombinant IGF-1 (rhIGF) for treatment of IGF-1 deficient short stature. This medication has not been studied in Crohn disease. The purpose of this study is to test the hypothesis that poor growth in Crohn disease is associated abnormal IGF-1 generation which leads to poor linear growth, decreased weight and osteoporosis and that replacement of IGF-1 with rhIGF will correct growth and improve bone density. To test our hypothesis we will recruit 20 patients with Crohn disease from our pediatric gastroenterology practice. Each will have been previously diagnosed with Crohn disease for a minimum of one year and will be studied at baseline and six month intervals for one year while on treatment with Increlex.

DETAILED DESCRIPTION:
1. Subjects. We will recruit 20 established Crohn patients from our gastroenterology (GI) referral practice at Nationwide Children's Hospital in Columbus, Ohio. Each will have previously undergone a complete diagnostic workup and classification of disease. Information on disease activity, location and behavior are routinely recorded at each follow up visit. Medical records will be assessed for this information. These patients will be followed every three months. All of these patients will be assigned to receive rhIGF therapy for 12 months and results will be compared to medical record data. We will recruit 10 per year.
2. Assessment of growth and IGF-1 generation. Each subject will undergo IGF-1 generation testing using standard published "high-dose: protocol and interpreted according to guidelines of Blum. Briefly, GH will be given as a one time per day subcutaneous injection in a dose of 0.05mg/kg/dy. IGF-1 will be measured at baseline and again after 7 days. Inadequate generation will be interpreted by an IGF-1 increase < 15 ng/dl after 7 days of GH. We will also measure baseline random GH and IGFBP-3 levels. The IGF-1, GH and IGFBP-3 levels will be measured by Esoterix laboratory (Calabasas Hills, CA). IGF-1 levels will also be measured every six months and with disease exacerbation. All patients will have a single radiological film of the left hand and wrist to determine bone age by Greulich and Pyle standards, and routine examination by the PI to determine Tanner staging.
3. Anthropometric measures. Patients will be seen every three months. At every visit, we will evaluate linear growth using a calibrated stadiometer and weight with a standardized scale. Longitudinal data will be used to calculate height and weight velocity. Height velocity will be annualized for each visit compared to baseline data. All growth information, including velocity will be converted to standard deviation scores (SDS, Z score) using GenenCalc (Genentech, San Francisco, CA).
4. Nutrition. To assess for low nutritional intake as the cause for poor growth (and low IGF-1 levels), each patient will complete a 3 day food journal at every visit and results will be assessed by Nutrition Pro software. We will evaluate our findings in both pubertal and prepubertal children. For this reason we will carefully measure Tanner stage as breast in girls and testicular volume in boys. We will measure testosterone levels in boys and estradiol in girls (Esoterix). Sex steroid levels will be correlated with Tanner staging and tempo of pubertal progression.
5. Treatment with rhIGF (Increlex, Tercica). Patients will be followed as above for 12 months while on Increlex therapy. Increlex (rhIGF) will be administered per the following schema: First 2 weeks: 40 mcg/kg BID; Weeks 3 and 4: 80 mcg/kg BID; Subsequent weeks: 120 mcg/kg BID. Each parent and patient will be carefully trained in injection technique by the same skilled personnel. Compliance will be assessed by having subjects return empty vials to the study site.
6. Bone mineral content and bone turnover. All subjects will undergo DXA scan (Lunar Prodigy) at baseline and every six months. Measurements will be compared to age- and gender- matched normals and converted to Z scores (www.bcm.edu/bodycomplab). To determine bone turnover, blood and urine will be collected at baseline and every six months. These labs will be run by Esoterix according to their methods: N-Telopeptides (reverse transcriptase PCR, urine), osteocalcin (double antibody RIA, blood), bone specific alkaline phosphatase activity (ICMA, blood), and deoxypyridinoline (ELISA, urine). Although the typical patient treated with GH demonstrates initial bone loss during the first six months, our group has documented improvement in bone mineral content within six months of starting GH therapy.
7. Cytokines. We will measure the cytokines TNF-α, IL-1, and IL-6 at the initiation of the study, at 6 months and 12 months. This will better help us understand the role of cytokines on disease course, activity, and the growth hormone axis.
8. Biomarkers for rhIGF-1 dosing efficacy. We will draw BL, 6 mos and 12 mos levels of IGF-1, IGFBP3 and ALS levels. The baseline level will be collected prior to the 1st dose of Increlex. At six months patients will be instructed to take their Increlex the morning of their visit and the sample will be drawn within 2 hours of dosing which will represent peak biomarker levels. The 12 month level will be obtained in the morning the day after the patient completes his/her final dose and will represent a trough level.
9. Measures of Disease Activity. At each protein turnover measure we will ask subjects to bring stool samples which will be evaluated for fecal calprotectin. We will complete the Pediatric Crohn Disease Activity Index (PCDAI), a reliable and valid index for disease activity in clinical research. Subjects will complete the IMPACT-III, a valid and reliable measure of quality of life in pediatric Crohn disease.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe Crohn Disease (PCDAI > 30)
* Chronological age 5-15 years old
* Tanner 1 - 3
* Bone age less than or equal to 13 in females and 14 in males

Exclusion Criteria:

* Identified infectious etiology
* Immunological disorder (excluding Crohn disease)
* Associated severe concomitant chronic illnesses (CF, liver failure, etc)

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2008-10; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dana S. Hardin, MD, Principal Investigator — The Research Institute at Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

REFERENCES:
- [Background] Cezard JP, Touati G, Alberti C, Hugot JP, Brinon C, Czernichow P. Growth in paediatric Crohn's disease. Horm Res. 2002;58 Suppl 1:11-5. doi: 10.1159/000064759. PMID 12373007
- [Background] Sentongo TA, Semeao EJ, Piccoli DA, Stallings VA, Zemel BS. Growth, body composition, and nutritional status in children and adolescents with Crohn's disease. J Pediatr Gastroenterol Nutr. 2000 Jul;31(1):33-40. doi: 10.1097/00005176-200007000-00009. PMID 10896068
- [Background] Hardin DS, Rice J, Doyle ME, Pavia A. Growth hormone improves protein catabolism and growth in prepubertal children with HIV infection. Clin Endocrinol (Oxf). 2005 Sep;63(3):259-62. doi: 10.1111/j.1365-2265.2005.02331.x. PMID 16117811
- [Background] Mauras N, George D, Evans J, Milov D, Abrams S, Rini A, Welch S, Haymond MW. Growth hormone has anabolic effects in glucocorticosteroid-dependent children with inflammatory bowel disease: a pilot study. Metabolism. 2002 Jan;51(1):127-35. doi: 10.1053/meta.2002.28972. PMID 11782884

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | rhIGF
Started | 3
Completed | 0
Not Completed | 3
Not completed — PI left and study terminated | 3

BASELINE CHARACTERISTICS:
Arm/Group | rhIGF
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.67 (2.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome Variable for the Monitoring Study (Baseline, Six Months and Disease Exacerbation) Will be Longitudinal Growth as Measured by Height Velocity
Time Frame: Six months and 1 year
Population: The PI left the institution suddenly and participant records stayed with the institution, so no analysis was able to be performed.
Arm/Group | rhIGF
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | rhIGF
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes